CLINICAL TRIAL: NCT05283226
Title: A Phase 2 Multicenter, Open-Label, Single-Arm Study to Evaluate the Safety and Efficacy of Oral NRC-2694-A in Combination With Paclitaxel in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma, Who Progressed on or After Immune Checkpoint Inhibitor Therapy
Brief Title: Study to Evaluate the Safety and Efficacy of Oral NRC-2694-A in Combination With Paclitaxel in Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma, Who Progressed on or After Immune Checkpoint Inhibitor Therapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NATCO Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAT2694US
Record Dates: First submitted 2022-02-08; First posted 2022-03-16 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma; Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma
Keywords: Carcinoma; Recurrent and/or Metastatic Cancer
MeSH Terms: conditions — Carcinoma | interventions — Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NRC-2694-A In Combination with paclitaxel (Experimental): Patients will receive NRC-2694-A 300 mg orally once daily and paclitaxel 175 mg/m² IV infusion over approximately 3 hours once in 21 days for 6 cycles or more.
  Interventions: Drug: NRC-2694-A; Drug: Paclitaxel

INTERVENTIONS:
Drug: NRC-2694-A — 300 mg orally once daily
Drug: Paclitaxel — 175 mg/m² IV infusion over approximately 3 hours

SUMMARY:
This is a Phase 2, open-label, multicenter, single-arm study of NRC-2694-A in combination with paclitaxel in patients with R/M HNSCC with progression on or after ICI therapy.

A total of approximately 46 male and female patients will be enrolled. This sample size is based on Simon's 2-stage design with historical control ORR of 30% and a target ORR of 50%.

DETAILED DESCRIPTION:
Patients with recurrent and/or metastatic unresectable Head and Neck Cancer have a poor prognosis and limited treatment options. Pembrolizumab and Nivolumab, both ICIs (Immune Checkpoint Inhibitors), are approved therapies for this condition. However, no approved treatment options exist for patients who progress on ICI therapies. Hence, there is an unmet medical need post-failure of ICI therapy. NRC-2694-A is an orally administered small-molecule tyrosine kinase inhibitor. It was discovered and developed by NATCO Pharma Ltd. NRC-2694-A demonstrated response in HNSCC patients in a Phase-I study as a monotherapy. This was further substantiated in a Phase-II study in combination with cisplatin/carboplatin and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and capable of understanding the written informed consent, provides signed and witnessed written informed consent, and agrees to comply with protocol requirements.
* Is male or female aged 18 years or older at the time of consent.
* Has histologically confirmed unresectable R/M HNSCC (oral cavity, oropharynx, hypopharynx, and larynx).
* Has documented progressive disease assessed by the principal investigator according to RECIST v1.1.
* Has a measurable lesion per RECIST v1.1.
* Has ECOG performance status score of ≤2.
* Must have progressed during or after receiving ICI therapy, such as pembrolizumab or nivolumab. Patients with prior immune-mediated reactions due to ICI therapies (eg, pembrolizumab or nivolumab) and who had recovered prior to study entry will also be eligible.
* Female patients of childbearing potential should have a negative urine test before enrollment. If the urine pregnancy test is positive or gives equivocal results, a serum pregnancy will be required for confirmation.
* Patients of reproductive age must use acceptable methods of contraception throughout the study period and for 30 days following the last dose of investigational product (see protocol for further guidance).
* During screening and at subsequent visits, the investigator should ensure adequate bone marrow reserve (neutrophil count ≥1500/mm3, platelet count ≥100,000/mm3, and hemoglobin level 8.0 g/dL), renal function (creatinine clearance ≥30 mL/min calculated by Cockcroft-Gault formula), liver function (total bilirubin level ≤1.5 × ULN [except patients with documented Gilbert's syndrome] and serum transaminase levels ≤2.5 × ULN or ≤5 × ULN for liver metastasis and/or obstructive jaundice).
* Must have completed a duration of at least two weeks after stopping ICI therapy/investigational therapy/salvage therapy and must have recovered to grade ≤1 from all toxicities due to such therapies.

Exclusion Criteria:

* Has cardiac, hepatic, endocrine, pulmonary, or autoimmune disease, interstitial lung disease, renal or psychiatric disorders, not controlled with therapy corresponding to the illness or a condition that contraindicates the use of a taxane or an EGFR inhibitor.
* Has Cirrhosis of liver at a level of Child-Pugh B (or worse).
* Has uncontrolled brain metastases. Patients are allowed if brain metastasis has been previously treated with surgery, whole brain irradiation, and/or stereotactic radiosurgery and are considered controlled (controlled by the dose ≤10 mg/day of prednisone or equivalent) at the time of the first dose of investigational product. Radiological evaluation of brain metastasis will be performed only if the patient has symptoms. For asymptomatic patients, brain imaging during screening is not required.
* Has baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTc interval >480 milliseconds [CTCAE Grade 1] using Fredericia's QT correction formula).
* Has a history of additional risk factors for Torsade de pointes (eg, heart failure, hypokalemia, family history of long QT syndrome).
* Has had prior cetuximab therapy for recurrent or metastatic disease. Note that cetuximab used concomitantly with radiotherapy or as an induction therapy is acceptable
* Has received any other EGFR-targeted therapies for recurrent or metastatic disease.
* Currently participating in any clinical trial or receiving investigational therapy on expanded access or compassionate basis.
* Has nasopharyngeal carcinomas or salivary gland cancers.
* Female patient who tested positive for pregnancy.
* Female patient who is breastfeeding or planning to become pregnant, or male patient planning to father a child within the duration of the study.
* Has tested positive for HIV, HBsAg, HCV antibody, or HCV RNA at screening. However, patients who test positive for HCV antibody, but negative for HCV RNA, will be allowed. In addition, patients with controlled HIV, chronic HBV on suppressive antiviral therapy, or a history of HCV infection status post-curative antiviral treatment with an HCV viral load below limit of quantification are permitted to participate (DHHS 2020).
* Has active infection requiring intravenous anti-infective therapy within 7 days prior to Day 1 Cycle 1 or is febrile due to infection.
* Has had major surgery within 4 weeks prior to screening.
* Administered a live attenuated vaccine within 4 weeks prior to Day 1 Cycle 1 or anticipation that such a live attenuated vaccine will be required during the study.
* Has known or suspected hypersensitivity to any components of the formulation used for this investigational product.
* Has concurrent disease or any clinically significant abnormality following the investigator's review of the screening physical examination findings, 12-lead ECG results, and clinical laboratory tests, which in the judgment of the investigator would interfere with the patient's participation in this study or evaluation of study results.
* Unable to come for study visits per schedule.
* Has current drug or alcohol abuse.
* Has received prior treatment with paclitaxel or docetaxel or any other drugs with taxane like mode of action for recurrent or metastatic or recurrent HNSCC. However, prior paclitaxel or docetaxel or any other drugs with taxane like mode of action as a component of a curatively-intended multimodality treatment for locally advanced HNSCC is permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2022-09-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To determine if NRC-2694-A administered orally in combination with paclitaxel demonstrates objective response in patients with R/M HNSCC, who have had radiological progression on or after treatment with ICI therapies like pembrolizumab or nivolumab | Baseline through approximately up to 24 weeks
  Objective response in terms of CR/PR per RECIST v1.1

SECONDARY OUTCOMES:
Progression-free survival | Baseline through approximately up to 24 weeks
  defined as the interval of time between the date of enrollment to the earliest date of disease progression, as determined by local radiologic assessment per RECIST v1.1, or death due to any cause, whichever occurs first
Overall survival | Baseline through approximately up to 24 weeks
  defined as the time from the date of enrollment to the date of death due to any cause
Duration of response | Baseline through approximately up to 24 weeks
  defined as the time from first confirmed objective response to disease progression
Clinical benefit response | Baseline through approximately up to 26 weeks
  defined as CR + PR + SD for ≥ 6 months
Number of adverse events | Baseline through approximately up to 24 weeks
Number of participants with abnormal physical examination findings | Baseline through approximately up to 24 weeks
  Symptom-directed physical examination will be conducted to evaluate skin rash, diarrhea, paresthesia, and dyspnea graded according to NCI CTCAE version 5.0.
Number of participants with abnormal vital signs | Baseline through approximately up to 24 weeks
  Clinically significant abnormal blood pressure, heart rate, respiratory rate, and oral body temperature graded according to NCI CTCAE version 5.0.
Assessing safety through ECOG (Eastern Cooperative Oncology Group) | Baseline through approximately up to 24 weeks
  The severity of the AE will be graded according to the NCI CTCAE version 5.0 (NCI Common Terminology Criteria for Adverse Events. The CTCAE displays Grades 1 through Grade 5 with the higher score as worse outcome)
Number of participants with abnormal clinical laboratory tests results | Baseline through approximately up to 24 weeks
  Clinically significant abnormal hematology, biochemistry, coagulation and urinalysis test results graded according to NCI CTCAE version 5.0.
Number of participants with abnormal ECGs (Electrocardiograms) | Baseline through approximately up to 24 weeks
  Clinically significant abnormal ECG findings will be graded per NCI CTCAE version 5.0.
Plasma PK parameters of NRC-2694-A measured via Cmax (Maximum plasma concentration) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via Tmax (time to reach the maximum plasma concentration) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via Ctrough (observed trough plasma concentration at the dosing interval tau) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via AUC0-t (area under the concentration-time curve from time zero to the time of last measurable concentration) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via AUC0-τ (area under the concentration-time curve from time zero to the dosing interval tau) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via CL/F (apparent clearance) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via Vz/F (apparent volume of distribution) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via Rac Cmax (accumulation ratio based on maximum plasma concentration) | Baseline through approximately up to 24 weeks
Plasma PK parameters of NRC-2694-A measured via Rac AUC (accumulation ratio based on area under the concentration-time curve) | Baseline through approximately up to 24 weeks

OTHER OUTCOMES:
To determine the association between NRC-2694-A activity and biomarkers in blood samples using Epidermal growth factor receptor status in EGFR (epidermal growth factor receptor) gene | Baseline through approximately up to 24 weeks
  as determined by NeoLAB® NGS platform biomarker assessment
To determine the association between NRC-2694-A activity and biomarkers in blood samples using downstream signaling in EGFR gene | Baseline through approximately up to 24 weeks
  as determined by NeoLAB® NGS platform biomarker assessment
To determine the association between NRC-2694-A activity and biomarkers in blood samples using mutations in EGFR gene | Baseline through approximately up to 24 weeks
  as determined by NeoLAB® NGS platform biomarker assessment

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Providence Medical Foundation -Fullerton, Fullerton, California
  - Los Angeles Hematology Oncology Medical Group, Los Angeles, California
  - Lynn Cancer Center, Boca Raton, Florida
  - Miami Cancer Center, Miami, Florida
  - Norton Cancer Institute - Downtown, Louisville, Kentucky
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - Washington University - Siteman Cancer Center, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Salib Oncology, Easton, Pennsylvania
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- India (3):
  - Daycare Angels under AOH, Mumbai, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - Basavatarakam Indo American Cancer Hospital & Research Institute, Hyderabad, Telangana

IPD SHARING:
Plan to Share IPD: No